CLINICAL TRIAL: NCT03642041
Title: Smoking Trajectory in Newly Diagnosis Lung Cancer Patients
Brief Title: Study of Smoking Trajectory in Newly Diagnosis Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Yang Chia Chen, Principal Investigator, National Defense Medical Center, Taiwan
Other Study IDs: TWNA-1042011
Record Dates: First submitted 2018-08-14; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Newly Diagnosed Lung Cancer; Smoking, Cigarette; Survival; Quality of Life
Keywords: Smoking; Lung cancer; Survival; Quality of life
MeSH Terms: conditions — Cigarette Smoking; Smoking; Lung Neoplasms | interventions — Smoking Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: smoking — smoking behavior

SUMMARY:
1. Understanding the smoking change patterns among the newly diagnosis lung cancer patients after cancer diagnosis.
2. Explore the related factors of the smoking change patterns.
3. The type of smoking trajectory impact on survival and quality of life.

DETAILED DESCRIPTION:
This was a prospective longitudinal design study. The investigators used the structure questionnaires to collect the data from a consecutive sample of newly diagnosed lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years old
* Newly diagnosed lung cancer
* Conscious clear and able to communicate
* Agreed to participate the study

Exclusion Criteria:

* Consciously confused
* Cognitive or psychotic disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2014-05-24 (Actual); Primary Completion 2017-07-22 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Changes From Baseline Smoking Behavior at 1,2,3,4,5,6 Months | baseline, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  Self-reported smoking during the last 30 days was a dichotomous variable.

SECONDARY OUTCOMES:
Changes From Baseline Quality of Life at 1,2,3,4,5,6 Months | baseline, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  Functional Assessment of Cancer Therapy-Lung, Version 4 (FACT-L v. 4) was a 36-item ordinal scale, five-point scale from 0 (not at all) to 4 (very much). There were 5 domains: Physical, social/family, emotional, and functional well-being; lung cancer subscale (symptoms, cognitive function, regret of smoking). Subscale scores added to obtain total score, with higher scores indicating better quality of life.
Proportion of participants with Overall Survival up to 2 years | follow up to one or two years
  survival